CLINICAL TRIAL: NCT06271889
Title: The Effect of Electro-fetal monıtorısıon Sound on Anxiety, paın and Postpartum
Brief Title: The Effect of Electro-fetal monıtorısıon Sound on Anxiety, paın and Postpartum Bonding at the First Phase of Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Assoc. Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.10.1.TKH.4.34.H.GP.0.01/330
Record Dates: First submitted 2021-12-02; First posted 2024-02-22 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Delivery Fear; Labor Pain; Maternal-Fetal Relations
Keywords: Fetal sound; Labor anxiety; Labor pain; Non Stress Test; Postpartum bonding
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: Randomized parallel controlled experimental design
Who Masked: Participant
Masking Description: Which of the participants is the control or intervention group will be selected by randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Control group pregnant women will be selected using randomization. their babies' fetal voice will not be listened.
- Intervention (Active Comparator): Pregnant women in the intervention group will be selected using randomization. the fetal voice of their babies will be listened to for about 3-5 minutes with a Non-stress Tester.
  Interventions: Device: Non-stress test

INTERVENTIONS:
Device: Non-stress test — It will be performed with the HUNTLEIGH brand BD4000XS-2 model NST device located at the maternity clinic to listen to the fetal heart sound, approximately min 3 max 5 min will be listened to. According to the studies conducted in the literature, the half-life of adrenaline in plasma is 3 minutes when an invasive/noninvasive intervention is performed on an adult individual. Therefore, the fetal heart rate will be listened to for 3 minutes (Dalal & Grujic; 2021; https://www.medicines.org.uk/emc/product/6284/smpc#gref https://www.ncbi.nlm.nih.gov/books/NBK482160 / )
  Arms: Intervention

SUMMARY:
University of Health Sciences, Istanbul Umraniye training and Research Hospital, Clinic of Obstetrics and gynecology, birth, maternity and Child Health Hospital, Aydın to the clinic, pregnant women, pregnant women in active labor act, and received acceptance to delivery to the fetal heart sound by existing tripped; fetal heart sounds of pregnant women, anxiety, pain and the birth in order to determine the effect of connecting the end of the level will be conducted. The study will guide midwives in reducing the anxiety or pain of pregnant women.

DETAILED DESCRIPTION:
Application of the Research: Informed voluntary consents will be obtained in written and oral form by giving the necessary information about the study to pregnant women before the application. The form will be signed ". Environmental stimuli before the procedure (noise, heat, light, touch, etc.) will be brought under control. Pregnant women admitted to the maternity hospital will be assigned to the intervention and control group using computer-aided randomization. Routine maintenance will be applied to both groups in the study. Anamnesis and blood are routinely taken from pregnant women admitted to the maternity unit within the scope of routine care in the institution where the research was conducted, and NST is connected by inserting an intravenous catheter. STAI and VAS will be filled in before the application to both groups of pregnant women. after application, the forms will be applied again at the beginning of the active phase (cervical opening 4-5 cm) and at the end (cervical opening 6-7 cm). In both groups; pulse, respiration and oxygen saturation will be evaluated with body temperature at the beginning of the active phase (cervical opening 4-5 cm) and at the end (cervical opening 6-7 cm) before and after the application. With decemberibel meter, the frequency range will be kept within the range of 30 dB-90 dB. Participants will be able to adjust the volume of their baby's voice at their own level. No noninvasive and invasive interventions will be applied to pregnant women in the intervention group during the application. If the control group is pregnant, only routine care will be performed. Both groups of pregnant women will be completed with STAI, VAS and the Postpartum Attachment scale before and after the application. The researcher should constantly monitor and evaluate the mother and fetus during the application process, and when discomfort develops, the procedure will be terminated and the clinical specialist physician will be informed.

ELIGIBILITY:
Inclusion Criteria:

* Who are december the age range of 18- 35,
* The least literate,
* Which is the primiparous,
* who is at the 38-42 week of gestation
* With a single pregnancy in the vertex position,
* Who does not have a systemic disease that will interfere with normal delivery (gestational diabetes, preeclampsia, etc.),
* Who is in the active phase of labor * Pregnant women who have agreed to participate in the study and received informed consent will be included in the study

Exclusion Criteria:

* 37. week 42. not between the weeks dec
* It is a multipart,
* Anyone who has any problems with communication,
* Who has ceased to be involved in the study,
* An unexpected complication develops (cesarean section of the pregnant woman, development of fetal distress in the fetus, etc.).

  * Oxytocin induction is applied Pregnant women who have been given pain medication (Aldolan, diazem) are

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2024-08-24 (Actual)

PRIMARY OUTCOMES:
VİSUAL ANALOG SCALE | immediately Before application
  Visual analog scale: The scoring system is between 0 and 10. 0 is considered as no pain, while 10 is considered as unbearable pain.
STATUS AND CONTINUOUS ANXIETY SCALE | immediately Before application
  The state anxiety scale consists of 20 statements. The state anxiety scale requires the individual to answer the feelings or behaviors experienced in the current situation by marking one of the options such as (1) Not at all, (2) A little, (3) A lot and (4) Completely according to the degree of severity.

OTHER OUTCOMES:
Postpartum Attachment Scale (PASAS): | In the first 24 hours postpartum after delivery
  Postpartum Attachment Scale (PASAS): It was developed by Brockington et al. (2001) to evaluate the mother's attachment to her baby in the postpartum period and to identify problems in the relationship between mother and baby. Turkish validity and reliability study was conducted (Yalçın et al, 2014). The scale, which was answered by mothers, consists of 25 questions and is a 6-point Likert-type scale defined as "always", "very often", "quite often", "sometimes", "rarely" and "never". 17 of the questions are calculated in reverse order. These questions are questions 2, 3, 5, 6, 7, 10, 12, 13, 14, 15, 17, 18, 19, 20, 21, 23, 24. High scores obtained from the scale indicate an increase in attachment problems.

CONTACTS AND LOCATIONS:
Overall Officials: Rojda BAYAR, PhD.Std., Study Chair — Istanbul Umraniye Training and Research Hospital; Ebru SAGIROGLU, PhD.Std., Principal Investigator — Uskudar University
Locations (1):
- Saglık Bilimleri Universitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lopez-Teijon M, Garcia-Faura A, Prats-Galino A. Fetal facial expression in response to intravaginal music emission. Ultrasound. 2015 Nov;23(4):216-223. doi: 10.1177/1742271X15609367. PMID 26539240
- [Result] Jelicic L, Jankovic S, Sovilj M, Adamovic T, Bogavac I, Gavrilovic A, Subotic M. Fetal Middle Cerebral Artery Pulsatility Index in No-Risk Pregnancies: Effects of Auditory Stimulation and Pregnancy Order. Int J Mol Sci. 2020 May 29;21(11):3855. doi: 10.3390/ijms21113855. PMID 32485789
- [Result] Aalbers S, Fusar-Poli L, Freeman RE, Spreen M, Ket JC, Vink AC, Maratos A, Crawford M, Chen XJ, Gold C. Music therapy for depression. Cochrane Database Syst Rev. 2017 Nov 16;11(11):CD004517. doi: 10.1002/14651858.CD004517.pub3. PMID 29144545
- [Result] Wulff V, Hepp P, Fehm T, Schaal NK. Music in Obstetrics: An Intervention Option to Reduce Tension, Pain and Stress. Geburtshilfe Frauenheilkd. 2017 Sep;77(9):967-975. doi: 10.1055/s-0043-118414. Epub 2017 Sep 25. PMID 28959060
- [Result] Corbijn van Willenswaard K, Lynn F, McNeill J, McQueen K, Dennis CL, Lobel M, Alderdice F. Music interventions to reduce stress and anxiety in pregnancy: a systematic review and meta-analysis. BMC Psychiatry. 2017 Jul 27;17(1):271. doi: 10.1186/s12888-017-1432-x. PMID 28750631
- [Result] Mahboubeh V, Masoumeh P, Zahra S. Comparison of vibro-acoustic stimulation and acupressure effects in nonstress test results and its parameters in pregnant women. Iran J Nurs Midwifery Res. 2013 Jul;18(4):266-71. PMID 24403920